CLINICAL TRIAL: NCT01153438
Title: Role of Endogenous Glucagon-like Peptide-1 (GLP-1) in Improved Glucose Tolerance After Two Different Types of Bariatric Surgery
Brief Title: Relationship Between Changes in Gut Hormones After Gastric Bypass and Gastric Banding and Improvements in Diabetes
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Marion L. Vetter, MD, RD, Principal Investigator, University of Pennsylvania
Other Study IDs: 810104
Record Dates: First submitted 2010-06-28; First posted 2010-06-30 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Type 2 Diabetes; Obesity; Bariatric Surgery
Keywords: Diabetes; Obesity; Bariatric surgery; Gut hormones; Glucagon like peptide 1; Insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Extra blood will be stored for the potential analysis of additional hormones.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Gastric bypass, Gastric banding

SUMMARY:
The purpose of this study is to see how hormones that control blood sugar change in response to two different weight loss surgeries (gastric bypass and gastric banding). We believe that changes in a hormone called glucagon-like peptide-1 (GLP-1) may account for the greater improvement in blood sugar after certain types of surgeries. GLP-1 makes the pancreas release insulin, a hormone that lowers blood sugar. The study will consist of one screening visit and three study visits in which the glucose response will be measured after drinking a liquid meal: 1) Visit 1 (2-3 weeks before surgery); 2) Visit 2 (after 10% of body weight is lost); and 3) Visit 3 (5-10 days after Visit 2). Hormone levels will be measured during the three study visits. To see if the improvement in blood sugar after surgery is due to changes in GLP-1, we will block its effect on insulin release by giving either salt water or a medication that blocks the activity of GLP-1 during the two visits that take place after surgery (Visits 2 and 3).

DETAILED DESCRIPTION:
Many diabetic patients who have Roux-en-Y gastric bypass (RYGB) have rapid improvements in their blood sugars within days of their surgery, even before they have lost much weight. It typically takes much longer for these improvements to occur after adjustable gastric banding (AGB), despite an equally low caloric intake. Changes in levels of hormones released by the small intestine as a consequence of the particular type of surgery may be an important factor in the rapid improvement of blood sugars. One of these hormones, glucagon-like peptide-1 (GLP-1), has an important effect on insulin secretion from the pancreas. This study seeks to determine whether changes in GLP-1 are responsible for the improvement in blood sugar after certain types of weight loss surgeries. In order to meet inclusion criteria, participants must have type 2 diabetes for less than 10 years and be approved by insurance to undergo RYGB or AGB at the Hospital of the University of Pennsylvania or Penn Presbyterian Medical Center. We will obtain several measurements of GLP-1 and other hormones that affect glucose levels during the three study visits: 1) Visit 1 (2-3 weeks before surgery); 2) Visit 2 (after 10% of body weight is lost); and 3) Visit 3 (5-10 days after Visit 2). To see if the improvement in blood sugar after surgery is due to changes in GLP-1, we will block its effect on insulin release by giving either salt water or a medication that blocks the activity of GLP-1 during the two visits that take place after surgery (Visits 2 and 3). Each visit will last for 4-6 hours and participants will be compensated for their time.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants age 18 years or older with a body mass index greater than >35 kg/m2 but less than <60 kg/m2 who undergo gastric bypass or gastric banding at the University of Pennsylvania.
* Type 2 diabetes (defined as a pre-existing diagnosis, the use of oral antidiabetic medications or insulin, or a fasting plasma glucose greater than or equal to > 126 mg/dl and confirmed by a oral glucose tolerance test)
* Ability to provide written informed consent

Exclusion Criteria:

* A diagnosis of type 1 diabetes
* Daily insulin requirement exceeding 1 unit/kg/d
* Poor preoperative glycemic control, as indicated by an HbA1c greater than 10.0%
* Duration of diabetes greater than> 10 years
* Pregnant women (or those who intend to become pregnant during the study period)
* Women who are currently breastfeeding
* Participants with moderate anemia (hemoglobin less than< 12 g/dl for men and less than< 11 g/dl for women)
* Use of medications known to affect weight, including chronic oral or inhaled glucocorticoid use and the use of certain psychiatric medications (olanzepine, risperidone, and lithium)
* history of any major active rheumatologic, pulmonary, dermatologic disease, or inflammatory conditions
* oral history of positive HIV status
* any major surgery in the past 3 months
* regular use of alcoholic beverages (greater than 7 drinks/week)
* prior reaction to human albumin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with type 2 diabetes who are medically approved and have insurance approval to undergo gastric bypass or gastric banding at the University of Pennsylvania.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2011-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
change in glucose tolerance after surgery (measured by glucose area under the curve) | after surgery when 10% of initial body weight is lost (expected 4 weeks after bypass and 12 weeks after banding)
  To compare change in glucose tolerance, independent of weight loss, between obese, diabetic participants who undergo gastric bypass or gastric banding.

SECONDARY OUTCOMES:
change in glucose tolerance before and after a GLP-1 receptor blocker is administered | after 10% of body weight is lost (expected 4 weeks after bypass and 12 weeks after banding)
  To determine if GLP-1 is responsible for improved glucose tolerance following gastric bypass.

CONTACTS AND LOCATIONS:
Overall Officials: Marion L Vetter, MD, RD, Principal Investigator — University of Pennsylvania
Locations (1):
- Center for Weight and Eating Disorders, University of Pennsylvania, Philadelphia, Pennsylvania, United States